CLINICAL TRIAL: NCT06395350
Title: Spire Health Remote Patient Monitor Human Factors Summative Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spire, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2019-337
Record Dates: First submitted 2019-09-27; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 17 adults for whom remote monitoring has been indicated by a health professional. At least 15 usable data points will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Spire Medical Health Tag (Other): Health Monitor Use
  Interventions: Device: Spire Health Monitor

INTERVENTIONS:
Device: Spire Health Monitor — Use of Health Monitor is Assessed

SUMMARY:
This usability validation testing protocol outlines the methods being used to demonstrate and gather evidence that the current design and user experience of the Spire Remote Patient Monitor are safe and effective for use by the people who are representative of the intended users under expected use conditions. This summative testing is the culmination of several preliminary analyses including a formative usability evaluation via Cognitive Expert Review Panel and is intended to assess the effectiveness of control measures put in place to reduce/eliminate use-related hazards or potential use errors.

DETAILED DESCRIPTION:
The summative testing will address user interactions with all components of the Spire Remote Patient Monitor related to tasks associated with the user group, including the Medical Health Tags, SpireHealth Mobile Application and Healthcare Provider Dashboard. This protocol specifies the required testing methods and associated acceptance criteria, as well as other information necessary to collect that evidence.

This human factors summative test is aimed to uncover the following:

* Determine if the final system design is safe and effective for use by the intended users in the intended use environment
* Investigation of any use errors related to risk observed
* To identify any potential new use errors relating to risk Background

Empirical activities in the form of a Cognitive Expert Review Panel was conducted to evaluate design iterations on critical tasks prior to summative testing. The results of these activities were used to improve UI design and inform analytical analyses such as task analysis, PCA analysis and use error analysis (DOC-75057 Use Error Analysis) This validation includes all Spire Remote Patient Monitor system interfaces associated with the primary consumer user groups.

The Spire Remote Patient Monitor that are the subject of this validation need to be supported by the following devices:

* SpireHealth Mobile Application running on a compatible smart phone (Apple iPhone or Android phone)
* Medical Health Tag device
* Spire Healthcare Provider Dashboard running in a browser on a personal computer

Prior to this summative testing there will be no training activities. Support and help are embedded within the app experience and Instructions for Use (IFU).

Seventeen (17) users will be recruited who comprise the single Spire Remote Patient Monitor user group: adults for whom remote monitoring has been indicated by a health professional. At least 15 usable data points will be collected. This sample size is based on the recommendation number of participants in IEC 62366: 2015, Part 1 and Part 2. The increased participant size is also to allow for cancellations and other test anomalies (e.g., equipment failures).

Session Description: 60 minutes, one-on-one session

Session Activities

1. Introduction and background questions: 5 minutes
2. Device in-use evaluation (observations and questions): 45 minutes
3. The final follow-up and closing: 10 minutes

The Facilitator's Script is allows for consistent interaction between the facilitators and the participants. As per the facilitator's discretion, any deviation to the exact script will be based on real-time responses to the session flow and responding the individual interaction. The script will have a list of questions specific to each scenario designed to help the facilitator/observer refine the information, to improve consistency of reporting, and assist the facilitator/observer in root cause analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must indicate that they are interested in using a smartphone and/or wearable fitness device for tracking their health
* High school degree or equivalent (e.g., GED) or less - at least 2
* Some college but no degree or associate degree - at least 4
* Age 22-49 - at least 5
* Age 50-65 - at least 5
* Age Over 65 - at least 2
* Near even split of men and women
* Almost never limited by my physical condition
* Rarely limited by my physical condition
* Occasionally limited by my physical condition
* Often limited by my physical condition
* Almost always limited by my physical condition
* Users with iPhone experience
* Smart Phone Savviness
* No more than 7 users who own use a wearable fitness device
* Wearable Fitness Device savviness

Exclusion Criteria:

* Participant currently works in tech industry
* Participant or a member of his/her household currently works for any company that develops, manufactures, or sells smartphones or smart wearable fitness devices
* Participant has participated in market or user research related to a medical device within the last 6 months and has participated in more than 2 in the last 3 years
* Participants are trained clinicians or healthcare providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Assess the participant's ability to perform essential tasks related to handling of device measured by Pass/Fail | 60 minutes
  Observational techniques will be used to assess the participant's ability to easily use various features on the device and discover whether user errors occur.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Medical Director for Clinimark LLC
Locations (1):
- Arthur Cabrera, MD., Louisville, Colorado, United States